CLINICAL TRIAL: NCT07022132
Title: Effects of Diaphragm Manual Therapy and Abdominal Hyporesive Exercises in Chronic Low Back Pain
Brief Title: Comparison of Physiotherapy Methods Applied To The Diaphragm In Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Humeyra Akil, Lecturer, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IMUFTR01
Record Dates: First submitted 2025-05-28; First posted 2025-06-15 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-07

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Conservative Treatment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diaphragmatic myofascial release (DMR) group (Active Comparator): This group will receive DMR in addition to conservative treatment consisting of stretching and strengthening exercises.
  Interventions: Other: Diaphragmatic myofascial release (DMR); Other: Conservative treatment
- Abdominal hypopressive exercise (AHE) group (Active Comparator): This group will receive AHE in addition to conservative treatment consisting of stretching and strengthening exercises.
  Interventions: Other: Abdominal hypopressive exercise (AHE); Other: Conservative treatment

INTERVENTIONS:
Other: Diaphragmatic myofascial release (DMR) — The physiotherapist, positioned on the head side of the supine patient, makes bilateral contact with the pisiform, hypothenar region and the underside of the 7th-10th costal cartilages with the last three fingers. During the inspiration phase, he/she pulls the contact points cephalically and slightly laterally with both hands, accompanying the elevation of the costae. During expiration, it deepens the contact towards the inner costal margin, maintaining resistance. In subsequent breathing cycles, it gradually increases the depth of contact inside the costal margin. The application is performed in 2 sets of 10 deep breaths with 1 minute between them.
  Arms: Diaphragmatic myofascial release (DMR) group
Other: Abdominal hypopressive exercise (AHE) — Each session consists of 6 hypopressive abdominal exercises with a 2-minute recovery period in between, and each exercise is repeated 3 times. This manoeuvre consists of expelling all air until the reserve volume is reached, then holding the breath (expiratory apnoea) and pulling the abdominal wall inwards and cranially by opening the costae without allowing air to enter. Exercises are performed in 6 different positions.
  Arms: Abdominal hypopressive exercise (AHE) group
Other: Conservative treatment — It consists of lumbar flexion and extension, stretching and strengthening exercises for the waist, back and abdominal region.

SUMMARY:
The aim of this study was to compare the effects of conservative treatment with diaphragmatic myofascial release (DMR) and abdominal hypopressive exercise (AHE) technique added to conservative treatment in chronic low back pain.

DETAILED DESCRIPTION:
Low back pain is one of the most common health problems in all societies and is a problem encountered by most individuals at some point in lifetime. Epidemiologic studies have shown that 70-80% of people complain of low back pain at some point in their lives. Low back pain, which ranks first in terms of chronic pain, causes pain, decreased normal joint movements, joint stiffness, loss of flexibility and activity limitations in individuals. These problems also cause difficulties in activities of daily living, decreased physical activity level, fear of movement and psychological stress, loss of work and performance, increased health expenditures and increased costs for employers.

Low back pain is often managed as a disease limited to isolated lumbar structures, but it often occurs in association with respiratory dysfunction, suggesting that low back pain is not an isolated musculoskeletal problem. Interestingly, the association between low back pain and respiratory disorders appears to be even stronger than the association with obesity and physical activity.

Due to its complex structure, the diaphragm has an important place in the postural chain. In addition to respiratory function, the diaphragm also plays an important role in stabilizing the spine during posture, balance and load-bearing activities, and therefore it is reasonable to assume that diaphragmatic dysfunction may also trigger low back problems.

Passive myofascial techniques are used to restore normal movement of the diaphragm and improve its function. It creates a greater pressure gradient between the thorax and abdomen and increases the expiratory phase. The biomechanical relationship between the diaphragm and other structures indicates that diaphragm techniques may have an effect on distal structures such as the Hamstring muscles, contributing to motor control and stabilization through activation of core stabilization muscles.

Training the muscles that form trunk stability can help improve low back pain. One of these training methods is the increasingly popular abdominal hypopressive exercises. The abdominal hypopressive exercise (AHE) technique was proposed by Marcel Caufriez in the 1980s for the treatment of pelvic floor disorders. The hypothesis of this method, which combines respiratory technique with abdominal contraction maneuvers, is that it relaxes the diaphragm, lowers intra-abdominal pressure and activates the abdominal muscles and pelvic floor simultaneously. Thus, it is suggested that urinary incontinence and pelvic organ prolapse can be reduced and that it can produce direct activation of the Transversus Abdominis muscle, which can strengthen the abdominal wall and stabilize the spine, increase the flexibility of the lumbar spine and Hamstring muscles, and reorganize body posture.

The aim of this study was to compare the effects of abdominal hypopressive exercise technique and myofascial diaphragm relaxation technique on pain, pressure pain threshold, functional status, range of motion, chest wall mobility, spinal mobility, flexibility and pelvic floor muscle activity in chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Experiencing low back pain for at least 12 weeks
* To be between the ages of 18-65

Exclusion Criteria:

* Pregnancy
* Severe osteoporosis
* Less than 1 year history of abdominal and/or thoracic surgery
* Having an additional disease such as severe coronary artery disease, uncontrolled hypertension, COPD that prevents exercise,
* Difficulty in co-operation
* History of malignancy
* History of lumbar spinal surgery
* Spondylolisthesis, scoliosis, other spinal deformities and congenital malformations
* Radiculopathy
* Systemic inflammatory diseases
* Corticosteroid injection in the last 3 months

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-08-10 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Pain intensity (Visual Analogue Scale) | 6 weeks
  The Visual Analogue Scale (VAS) will be used to assess the level of pain at rest and during movement. The VAS is a self-reported scale consisting of a horizontal or vertical line, usually 100 millimetres long, with two verbal descriptors indicating pain status at the extremes. The patient is asked to indicate where on this line his/her condition fits by drawing a line, putting a dot or pointing.

SECONDARY OUTCOMES:
Hamstring flexibility (The Active Knee Extension Test) | 6 weeks
  The Active Knee Extension Test (AKET) starts in the supine position with the hip and knee in 90° flexion. In this position and with the axis of the goniometer placed on the lateral condyle of the femur, the subject is asked to perform knee extension without changing the flexion of the hip and avoiding pelvic movements. The angle remaining for full extension of the knee reflects the degree of hamstring shortening.
Chest wall mobility (a tape measure) | 6 weeks
  Chest wall mobility will be measured with a tape measure during full inspiration and full expiration.
Pelvic floor muscle activity | 6 weeks
  Pelvic floor muscle activity will be evaluated by surface EMG.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Hümeyra Akıl, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No